CLINICAL TRIAL: NCT00187434
Title: A Randomized Control Trial Comparing Two Methods of Delivering Continuous Positive Airway Pressure (CPAP), Infant Flow System CPAP and Bubble CPAP, in Supporting Successful Extubation of Infants of Birth Weights Less Than or Equal to 1500 Grams at Birth (C2CPAP)
Brief Title: Comparison of Two Methods of Continuous Positive Airway Pressure (CPAP) to Support Successful Extubation of Infants of Birth Weights ≤ 1500 Grams (C2CPAP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Lung Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240-2003
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2007-01-23 (Estimated); Status verified 2005-09

CONDITIONS: Premature Birth; Respiratory Insufficiency
Keywords: premature infant; supporting extubation
MeSH Terms: conditions — Premature Birth; Respiratory Insufficiency

INTERVENTIONS:
Device: Infant Flow System
Device: Bubble CPAP

SUMMARY:
Continuous positive airway pressure (CPAP) has been used successfully to promote extubation in the premature infant population. The two methods of CPAP to be examined are currently used by many institutions, yet no study has compared these methods to determine which is better in the population of newborns < 1500 grams (birth weight) at supporting extubation. This randomised controlled study will examine two types of CPAP: the Infant Flow System and the Bubble CPAP. This randomised controlled, single site, clinical study is to determine whether the Bubble CPAP or the Infant Flow System (IFS) CPAP is more effective at supporting the extubation in infants of birth weights < 1500 grams. Seventy-six infants will be randomised, immediately prior to extubation, to IFS or Bubble CPAP of 5 cmH2O. The primary outcome is successful extubation, defined as not reaching failure criteria for the 7 days post-extubation. Failure criteria are defined as pH < 7.25 and PCO2 > 65 mmHg or a sustained increase in FiO2 of 0.15.

DETAILED DESCRIPTION:
Background: Continuous Positive Airway Pressure (CPAP) has been used successfully to promote extubation in the premature infant population (Davis & Henderson-Smart, 2002). The two methods of CPAP to be examined are used by many institutions, yet no study has compared these methods to determine which is better in the population of newborns < 1500 grams (birth weight) at supporting extubation. This study may have cost savings implications. If bubble CPAP is shown to be as effective in this application neonatal intensive care units (NICUs) will have a more affordable option of providing effective CPAP.

Methods: This randomised controlled, single site, clinical study is to determine if Bubble CPAP or Infant Flow System (IFS) CPAP is more effective at supporting extubation in infants of birth weights < 1500 grams. Seventy-six infants will be randomised immediately prior to extubation to IFS or Bubble CPAP of 5 cmH2O. The primary outcome is successful extubation, defined as not reaching failure criteria for the 7 days post-extubation. Failure criteria are defined as pH < 7.25 and PCO2 > 65 mmHg or a sustained increase in FiO2 of 0.15.

Participants: Parents/guardians of eligible infants will be approached and given information regarding the study, and any questions answered. They will then be allowed to consider study participation in private. The recruiter will return at an agreed time and informed consent will be obtained from those agreeing to participate. Parents will be approached in accordance with the guidelines of the NICU @ SWCHSC. Infants are eligible if birth weight < 1500 grams, are to be extubated to CPAP and have no known airway anomalies, or suspected genetic anomalies.

Analysis: Multiple ANOVA analysis will be used for continuous variables, chi-square for categorical variables, including primary outcome.

Conclusion: The results of this study will determine which method of CPAP is the best method of supporting extubation in the < 1500 g infant.

ELIGIBILITY:
Inclusion Criteria:

* Intubated infant
* ≤ 1500 grams at birth
* Decision to extubate to CPAP made by the clinical team
* Written informed consent obtained

Exclusion Criteria:

* Have known airway anomalies
* Have grade III or IV or periventricular leukomalacia
* Have known or suspected genetic syndromes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76
Dates: Start 2003-09

PRIMARY OUTCOMES:
failure of extubation as defined by the following: pH < 7.25 and PCO2 > 65 (or an increase of 15 mmHg from pre-extubation), a sustained (> 1 hour) increase in FiO2 of .15 (as compared to pre-extubation) or significant apno

SECONDARY OUTCOMES:
reintubation
length of time in days on CPAP
corrected gestational age at cessation of CPAP
average weight gain on CPAP
assessment of pain will

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn D Hyndman, Principal Investigator — Sunnybrook & Women's College Health Sciences Centre
Locations (1):
- Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ho JJ, Zakarija-Grkovic I, Lok JW, Lim E, Subramaniam P, Leong JJ. Continuous positive airway pressure (CPAP) for apnoea of prematurity. Cochrane Database Syst Rev. 2023 Jul 18;7(7):CD013660. doi: 10.1002/14651858.CD013660.pub2. PMID 37481707